CLINICAL TRIAL: NCT07391722
Title: A Multicentre, Randomized, Double-Blind, Placebo-controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of DNV001 Injection at Different Dosages in Patients With Primary Hypercholesterolaemia or Mixed Hyperlipidaemia and Elevated Low Density Lipoprotein Cholesterol (LDL-C) Inadequate
Brief Title: DNV001 Injection in Patients With Hypercholesterolemia
Acronym: DNV001
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hangzhou Dinovate Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DNV001-201; 2025LP01037 (Other: NMPA)
Record Dates: First submitted 2025-12-14; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Primary Hypercholesterolemia
Keywords: DNV001; PCSK9 inhibitor; LDL-C; Hypercholesterolemia; Mixed dyslipidemia; Randomized controlled trial
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel-group design with four active dose arms and a shared placebo control within each arm (4:1 randomization per arm).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study where both the participants and the investigators (including site personnel involved in treatment administration and clinical evaluation) are masked to treatment assignment. The placebo is matched in packaging, and administration to maintain blinding. The sponsor's clinical and monitoring staff are also masked. Unblinding may occur only in medical emergencies per the study protocol. An independent unblinded pharmacist,nurses or designated staff at each site will handle randomization and drug dispensing to maintain allocation concealment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- DNV001-50 mg (Experimental): Participants receive DNV001 50 mg via subcutaneous injection at Day 1, Week 12, and Week 36, while continuing their stable background statin therapy.
  Interventions: Biological: DNV001 Injection
- DNV001-150 mg (Experimental): Participants receive DNV001 150 mg via subcutaneous injection at Day 1, Week 12, and Week
  Interventions: Biological: DNV001 Injection
- DNV001-300-1 mg (Experimental): Participants receive DNV001 300 mg via subcutaneous injection at Day 1, Week 12, and Week 36, while continuing their stable background statin therapy.
  Interventions: Biological: DNV001 Injection
- DNV001-300-2 mg (Experimental): Participants receive DNV001 300 mg via subcutaneous injection at Day 1 and Week 24 (only two doses), while continuing their stable background statin therapy.
  Interventions: Biological: DNV001 Injection
- Placebo (Placebo Comparator): Participants receive matching placebo via subcutaneous injection according to the schedule of the DNV001 dose group to which they are randomized (e.g., at Day 1, Week 12, and Week 36 for the 50 mg, 150 mg, and 300 mg-1 groups; or at Day 1 and Week 24 for the 300 mg-2 group), while continuing their stable background statin therapy.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: DNV001 Injection — DNV001 is a human monoclonal antibody targeting PCSK9 (proprotein convertase subtilisin/kexin type 9), administered as a sterile solution for subcutaneous injection. It is supplied in a 1.5 mL type I borosilicate glass vial with a concentration of 200 mg/mL (300 mg per vial). The product should be stored at or below 25°C and must not be frozen
  Arms: DNV001-150 mg; DNV001-300-1 mg; DNV001-300-2 mg; DNV001-50 mg
Biological: Placebo — Matching placebo for DNV001 injection. It is identical in appearance, packaging, and administration route to the active drug, but does not contain the active pharmaceutical ingredient. Supplied in a 1.5 mL vial for subcutaneous injection and stored under the same conditions (≤25°C, do not freeze).
  Arms: Placebo

SUMMARY:
This is a Phase II clinical study to evaluate the effectiveness and safety of different doses of DNV001 injection in patients with primary hypercholesterolemia or mixed dyslipidemia who have not achieved adequate control of low-density lipoprotein cholesterol (LDL-C) despite statin therapy.

The study will enroll approximately 120 participants and will be conducted at 10-15 centers in China. Participants will be randomly assigned to one of four dose groups (50 mg, 150 mg, 300 mg-1, or 300 mg-2) or placebo, administered as subcutaneous injections. The study includes a 2-week screening period, a 4-week run-in period, a 36-week double-blind treatment period, and a 12-week follow-up period, for a total of up to 54 weeks.

The main goal is to see how much DNV001 lowers LDL-C levels after 24 weeks of treatment. The study will also look at long-term effectiveness, safety, how the body processes the drug, and whether it causes an immune response.

All participants will continue taking their stable dose of statin medication throughout the study.

DETAILED DESCRIPTION:
Study Title:

A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of Different Doses of DNV001 Injection in Patients with Primary Hypercholesterolemia or Mixed Dyslipidemia with Elevated LDL-C Despite Statin Therapy.

Sponsor:

Hangzhou Dinovate Biotech Co., Ltd.

Protocol Number:

DNV001-201

Phase:

Phase II

Study Design:

This is a randomized, double-blind, multicenter, placebo-controlled study. Eligible participants will be assigned in a 1:1:1:1 ratio to one of four dose groups: 50 mg, 150 mg, 300 mg-1, or 300 mg-2. Within each dose group, participants will be further randomized 4:1 to receive either DNV001 or placebo. Each dose group will include 24 participants receiving active drug and 6 receiving placebo, for a total of approximately 96 active and 24 placebo participants.

Study Duration:

Each participant will be involved for up to 54 weeks, including:

* Screening: 2 weeks
* Run-in: 4 weeks
* Double-blind treatment: 36 weeks
* Follow-up: 12 weeks

Key Eligibility Criteria:

Inclusion:

* Adults ≥18 years with primary hypercholesterolemia or mixed dyslipidemia
* Inadequate LDL-C control despite stable statin therapy
* Fasting LDL-C ≥70 mg/dL (with ASCVD history) or ≥100 mg/dL (without ASCVD history)
* Fasting triglycerides ≤400 mg/dL
* Willing to comply with study visits and lifestyle/dietary guidelines

Exclusion:

* Homozygous familial hypercholesterolemia
* Recent major cardiovascular event or procedure
* Uncontrolled hypertension, diabetes, or thyroid disease
* Significant liver, kidney, or heart disease
* Use of other lipid-lowering therapies (except stable statins)
* Recent participation in another clinical trial

Endpoints:

Primary:

· Percent change in LDL-C from baseline at Week 24.

Secondary:

* Percent change in LDL-C at other timepoints up to Week 48
* Proportion of participants achieving LDL-C reduction ≥50%, LDL-C <70 mg/dL, etc.
* Safety (adverse events, lab abnormalities, ECG, vital signs)
* Pharmacodynamics (PCSK9, lipids, lipoproteins)
* Pharmacokinetics (Cmax, Tmax, AUC)
* Immunogenicity (anti-drug antibodies)

Intervention:

DNV001 or matching placebo will be administered subcutaneously in the abdomen, upper arm, or thigh. Dosing schedules vary by group (e.g., 50 mg group: doses at Day 1, Week 12, Week 36; 300 mg-2 group: Day 1 and Week 24).

Statistical Methods:

Analyses will be performed on the Full Analysis Set, Per Protocol Set, and Safety Set. The primary endpoint will be analyzed using a mixed model for repeated measures. Safety and other endpoints will be summarized descriptively.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria to be eligible for inclusion in this study:

  1. Male or female, aged ≥18 years at the time of signing the informed consent form;
  2. Diagnosed with primary hypercholesterolaemia or mixed hyperlipidaemia at screening; have been receiving statin therapy prior to screening; and agree to maintain stable statin therapy (i.e., no change in type or dosage, except for safety reasons) throughout the study;
  3. Fasting LDL-C levels at both the screening and run-in periods must meet the following criteria, as tested by a local laboratory: For subjects with a documented history of ASCVD, fasting LDL-C must be ≥ 70 mg/dL (1.8 mmol/L). For subjects without a documented history of ASCVD, fasting LDL-C must be ≥ 100 mg/dL (2.6 mmol/L);
  4. Fasting TG ≤ 4.52 mmol/L (400 mg/dL), as tested by a local laboratory, at both the screening and run-in periods;
  5. Understand the study procedures and methods, voluntarily agree to participate in this study, be willing to comply with the visit schedule and protocol requirements, and provide written informed consent;
  6. Be willing to adhere to the lifestyle requirements specified in the study protocol (including diet and physical activity level) during the study;
  7. Female subjects of childbearing potential (WOCBP) and male subjects who have not undergone vasectomy must agree to use a reliable method of contraception during the study and 6 months after study completion or discontinuation; female subjects of childbearing potential must present negative for blood human chorionic gonadotropin (hCG) pregnancy test result at the screening visit and the baseline visit prior to the first dose; male subjects must not donate sperm during the study and for 6 months after study completion or discontinuation.

Exclusion Criteria:

* Subjects who meet any of the following criteria will not be enrolled in the study:

  1. Diagnosed with homozygous familial hypercholesterolaemia prior to screening;
  2. Assessed as having an ultra-high risk for overall ASCVD at screening and have undergone percutaneous coronary intervention within 1 year prior to screening;
  3. Have other diseases that significantly affect blood lipid levels (such as nephrotic syndrome, severe liver diseases) or have dyslipidemia due to other secondary causes (such as drug-induced dyslipidemia);
  4. History of allergy to drugs or foods (two or more), or a history of specific allergic diseases (such as asthma, urticaria, eczematous dermatitis, etc.), or known allergy to any active ingredient or excipient of the investigational product;
  5. History of malignancy within the past 5 years (except for cured basal cell carcinoma of the skin, etc.), or currently being evaluated for a potential malignancy;
  6. Office blood pressure measurement during the screening and run-in periods: systolic blood pressure (SBP) ≥ 180 mmHg or diastolic blood pressure (DBP) ≥ 110 mmHg (a repeat measurement is permitted, which must be completed on the same day, and no pharmacological intervention is allowed before the repeat measurement);
  7. History of serious cardiovascular or cerebrovascular diseases (such as hypertensive encephalopathy, acute stroke, transient ischemic attack, acute myocardial infarction, severe arrhythmia), or severe aortic and/or peripheral vascular diseases (such as abdominal aortic aneurysm, lower limb arteriosclerosis obliterans), or presence of indications for surgical intervention within 6 months prior to screening or during the run-in period;
  8. Underwent major surgery within 6 months prior to screening or during the run-in period, or plan to undergo major surgery during the study period;
  9. History of New York Heart Association (NYHA) class III-IV heart failure, with a left ventricular ejection fraction (LVEF) < 40% at screening or run-in period;
  10. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 (calculated using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation) at screening or run-in period;
  11. Presence of severe thyroid disease (except for those on stable thyroxine replacement therapy or anti-thyroid drug therapy for at least 6 months prior to screening);
  12. Meet any of the following conditions in laboratory tests at screening or run-in period:

      * Thyroid stimulating hormone (TSH) > 1.5 × upper limit of normal (ULN) or < 1.0 × ULN;
      * Creatine kinase (CK) > 3×ULN;
      * Alanine aminotransferase (ALT), aspartate aminotransferase (AST) >2×ULN;
      * Total bilirubin (TBIL): 1.5×ULN.
  13. QT/QTcF interval prolongation (≥ 450 ms for male subjects or ≥ 470 ms for female subjects) at screening or run-in period;
  14. Positive result for either human immunodeficiency virus antibody (HIV-Ab) or treponema pallidum antibody (TP-Ab); positive for hepatitis B surface antigen (HBsAg) with hepatitis B virus load (HBV-DNA) exceeding the upper limit of the local laboratory reference range; or positive for hepatitis C virus antibody (HCV-Ab) with hepatitis C virus load (HCV-RNA) exceeding the upper limit of the local laboratory reference range;
  15. Poorly controlled type 1 or type 2 diabetes mellitus during the screening or run-in period, defined as glycosylated hemoglobin (HbA1c) > 8.5%; or newly diagnosed type 2 diabetes mellitus within 3 months prior to screening;
  16. History of drug abuse, including repeated high-dose use of dependence-inducing drugs or substances unrelated to medical purposes, including addictive or habitual drugs that cause physical or psychological dependence;
  17. History of alcohol abuse, defined as consumption of more than 14 standard units of alcohol per week within the past 6 months (one standard unit equals 14 g of pure alcohol, e.g., 360 mL beer, 45 mL spirits [≥ 40% alcohol], or 150 mL wine);
  18. History of blood donation within 3 months prior to screening or during the run-in period or blood loss ≥ 400 mL within 6 months prior to randomization (except blood loss due to menstruation);
  19. Weight change (gain or loss) of ≥ 10% within 3 months prior to screening;
  20. Received any medication or health product, other than the investigational product and stable-dose statin background therapy, that affects blood lipid levels within 4 weeks or 5 drug half-lives (whichever is longer) prior to randomization, including but not limited to: other statins (except stable statins), ezetimibe and similar agents (e.g., hybutimibe), fibrates, fish oil, niacin, bile acid sequestrants (e.g., cholestyramine), obesity treatment drugs, soluble fiber supplements, plant sterol-enriched margarines, glucagon like peptide-1 (GLP-1) receptor agonists, traditional Chinese medicines or Chinese patent medicines with lipid-lowering effect;
  21. Received monoclonal antibody PCSK9 inhibitors within 180 days prior to randomization, or small interfering RNA (siRNA)-based PCSK9 inhibitors (e.g., inclisiran) within 12 months prior to randomization;
  22. Use of drugs or foods contraindicated with statins prior to screening or randomization, without a discontinuation period of at least 5 drug half-lives, e.g., cyclosporine;
  23. Received systemic glucocorticoids (e.g., prednisone > 15 mg/d or other equivalent doses), thiazide diuretics, β-blockers, and other medications that may affect blood lipid levels within 4 weeks or 5 drug half-lives (whichever is longer) prior to screening or randomization, except for stable, low-dose use deemed by the investigator not to affect blood lipids;
  24. Participated in any clinical study and received the investigational drug/device within 3 months prior to screening or 5 half lives (whichever is longer) of the investigational drug, or before randomization, or planning to participate in any other clinical study during the study period;
  25. Pregnant or lactating women, or women of childbearing potential, male participants who plan to conceive (including sperm and egg donation) during the study period and/or who do not agree to use effective contraception;
  26. Any other conditions that, at the discretion of the investigator, would make the subject unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility for participation is based on biological sex (male or female), as defined in the study protocol. All individuals who meet the medical eligibility criteria, regardless of their gender identity, are welcome to participate.
Enrollment: 120 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of DNV001 in subjects with primary hypercholesterolaemia or mixed hyperlipidaemia with elevated LDL-C levels | Baseline to Week 24
  Percent change from baseline in LDL-C levels at Week 24 (W24).

SECONDARY OUTCOMES:
To evaluate other efficacy measures of DNV001 in subjects with primary hypercholesterolaemia or mixed hyperlipidaemia with elevated LDL-C levels | Baseline to Week 48
  ● Key secondary endpoints: Percent change from baseline in LDL-C levels at Week 48 (W48);
To evaluate other efficacy measures of DNV001 in subjects with primary hypercholesterolaemia or mixed hyperlipidaemia with elevated LDL-C levels | Baseline to Week 48
  ● Percent change from baseline in LDL-C levels at W2, W4, W8, W12, W14, W16, W20, W28, W32, W36, W40, W44;
To evaluate other efficacy measures of DNV001 in subjects with primary hypercholesterolaemia or mixed hyperlipidaemia with elevated LDL-C levels | Baseline to Week 48
  ● Proportion of subjects whose LDL-C levels are restored to 80% or more of baseline levels at W24, W36, and W48;
To evaluate other efficacy measures of DNV001 in subjects with primary hypercholesterolaemia or mixed hyperlipidaemia with elevated LDL-C levels | Baseline to Week 48
  ● Proportion of subjects whose LDL-C levels have decreased by ≥ 50% from baseline at W24, W36, and W48;
To evaluate other efficacy measures of DNV001 in subjects with primary hypercholesterolaemia or mixed hyperlipidaemia with elevated LDL-C levels | Baseline to Week 48
  ● Proportions of subjects with LDL-C < 0.65 mmol/L (25 mg/dL), < 1.3 mmol/L (50 mg/dL), < 1.8 mmol/L (70 mg/dL), and < 2.6 mmol/L (100 mg/dL) at W24, W36, and W48;
To evaluate other efficacy measures of DNV001 in subjects with primary hypercholesterolaemia or mixed hyperlipidaemia with elevated LDL-C levels | Baseline to Week 48
  ● Proportion of subjects achieving the LDL-C target according to atherosclerotic cardiovascular disease (ASCVD) risks categories at W24, W28, W32, W36, W40, W44, and W48.
To evaluate the safety of DNV001 in subjects with primary hypercholesterolaemia or mixed hyperlipidaemia with elevated LDL-C levels | Baseline to Week 48
  ● The incidence and severity of adverse events (AEs) and serious adverse events (SAEs) during the study;
To evaluate the safety of DNV001 in subjects with primary hypercholesterolaemia or mixed hyperlipidaemia with elevated LDL-C levels | Baseline to Week 48
  ● Abnormal changes in laboratory tests, electrocardiograms (ECGs), vital signs, physical examinations, etc. during the study.
To characterize the pharmacodynamics (PD) of DNV001 in subjects with primary hypercholesterolaemia or mixed hyperlipidaemia with elevated LDL-C levels | Baseline to Week 48
  ● Changes from baseline in the levels of PCSK9 and other lipid levels, lipoprotein, and apolipoprotein (including triglycerides [TG], total cholesterol [TC], high density lipoprotein cholesterol [HDL-C], apolipoprotein A1 [ApoA1], apolipoprotein B [ApoB], small dense low density lipoprotein [sdLDL-C], and lipoprotein(a) [Lp(a)]) at each assessment time point.
To characterize the pharmacokinetics (PK) of DNV001 in subjects with primary hypercholesterolaemia or mixed hyperlipidaemia with elevated LDL-C levels | Baseline to Week 48
  ● Analysis of blood concentrations and PK parameters of DNV001 (including peak concentration [Cmax] at specific treatment time points in individuals and groups.
To characterize the pharmacokinetics (PK) of DNV001 in subjects with primary hypercholesterolaemia or mixed hyperlipidaemia with elevated LDL-C levels | Baseline to Week 48
  ● Analysis of blood concentrations and PK parameters of DNV001 including time to peak concentration [Tmax] at specific treatment time points in individuals and groups.
To characterize the pharmacokinetics (PK) of DNV001 in subjects with primary hypercholesterolaemia or mixed hyperlipidaemia with elevated LDL-C levels | Baseline to Week 48
  ● Analysis of blood concentrations and PK parameters of DNV001 including area under the time-concentration curve [AUC], etc.) at specific treatment time points in individuals and groups.
To evaluate the immunogenicity of DNV001. | Baseline to Week 48
  ● Incidence of anti-drug antibodies (ADA) (including the positive rate and antibody titers of ADA).

OTHER OUTCOMES:
To evaluate the effect of DNV001 on the steady-state blood concentrations of statins (atorvastatin) in subjects with primary hypercholesterolaemia or mixed hyperlipidaemia with elevated LDL-C levels | Baseline to Week 48
  ● Analysis of steady-state blood concentrations of statins (atorvastatin) at specific treatment time points in individuals and groups.

IPD SHARING:
Plan to Share IPD: Undecided
A decision regarding sharing of de-identified individual participant data (IPD) has not yet been made by the sponsor. Any future plan for data sharing will consider factors such as the completion of the study, publication of primary results, and regulatory approvals. This record will be updated if a sharing plan is established.